CLINICAL TRIAL: NCT00341354
Title: Evaluation of Silver-Sulfadiazine Tracheal Tubes / Mucus Shaver in Intubated Patients Expected to Have a Prolonged Mechanical Ventilation
Brief Title: Coated Endotracheal Tube and Mucus Shaver to Prevent Hospital-Acquired Infections
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 999906087; 06-H-N087
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-09-06

CONDITIONS: Infection
Keywords: Pneumonia; Bacterial Infection; Nosocomial Infection; Trachea; Biofilm; Mucus Shaver
MeSH Terms: conditions — Infections; Pneumonia; Bacterial Infections; Cross Infection; Tracheal Diseases

INTERVENTIONS:
Behavioral: Prolonged Mechanical Ventilation

SUMMARY:
This study, conducted at the San Gerardo Hospital in Milan, Italy, will examine whether a bacteriocidal-coated endotracheal tube (breathing tube) cleaned with a device called a Mucus Shaver is safe and effective in preventing hospital-acquired infections in patients who require prolonged mechanical ventilation in an intensive care unit (ICU).

Pneumonia is the most frequent hospital-acquired infection in the ICU; its development is likely related to the use of a breathing tube. The tube is placed in the patient's trachea (windpipe) to assist breathing during and after an operation. Currently, breathing tubes in intubated patients are cleaned with a suction catheter that draws out secretions that accumulate in the tube. This method does not clean the tube completely, however, and within a few hours after the breathing tube is placed, bacteria may begin to grow inside the tube. Over time, as the patient breathes in and out through the tube, the bacteria may break free and enter the lungs, possibly causing pneumonia. In addition, the growth of bacteria in the tube decreases the size of the airway passage, making it more difficult to keep air moving in and out of the lungs.

Previous studies have shown that breathing tubes coated with silver-sulfadiazine prevented bacterial growth in the patient's airways and that use of the Mucus Shaver prevented accumulation of secretions in the lumen of the breathing tube, keeping the tube open. This study will determine if use of the coated tube and Mucus Shaver in patients requiring prolonged mechanical ventilation is safe and if it can reduce bacterial growth, the length of intubation and mechanical ventilation, the occurrence of pneumonia and the length of time in ICU and hospital.

Patients at San Gerardo Hospital who are 18 and older, who expect to have a breathing tube in place for more than 48 hours, and who are not allergic to silver-sulfadiazine may be eligible for this study.

Participants are randomly assigned to have either a standard breathing tube and standard cleaning or a coated tube cleaned with a Mucus Shaver. At intubation, a sample of secretions is collected from the mouth, the lumen of the breathing tube, and the airways. The lumen of the breathing tube is then cultured every day. When the tube is removed, or on the eighth day of intubation, a sample of secretions is collected from the mouth, the lumen of the breathing tube, and the airways. After the tube is removed, it is examined for biological and microscopic analysis.

DETAILED DESCRIPTION:
Pneumonia is the most frequent hospital-acquired infection in the intensive care unit, having a significant mortality, morbidity and cost. It occurs frequently in patients who are intubated and on a ventilator. In two phase I/II clinical studies, we tested endotracheal tubes (ETT), internally coated with bacteriocidal agents, and the Mucus Shaver, which removes material from the inside of the endotracheal tube. We showed 1) no adverse events, 2) that coating the inner wall of the ETT with silver-sulfadiazine significantly reduced bacterial colonization of the ETT; and 3) the Mucus Shaver cleans the lumen, leaving the entire endotracheal tube free of secretions, and maintains the lumen diameter. In this study, to evaluate the safety and effectiveness of the Mucus Shaver with the coated ETT, we propose to conduct a randomized trial in intubated patients on prolonged mechanical ventilation.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Males and females greater than 18 years old;
  2. Patients who are expected to be intubated and mechanically ventilated for greater than 48 hours;
  3. Patients who require an endotracheal tube with an internal diameter of 7.5 mm or 8.0 mm.

EXCLUSION CRITERIA:

1. Males and females less than 18 years old;
2. Patients who are expected to be intubated for less than 48 hours;
3. Patients who are allergic to silver-sulfadiazine;
4. Patients who require an internal diameter of an endotracheal tube less than 7.5 mm or greater than 8.0 mm;
5. Patients who do not tolerate disconnection from the ventilator:

   * Hemodynamically unstable;
   * Severe ARDS: PaO2/FiO2 less than or equal to 200 at PEEP less than or equal to 5 cmH20.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 2006-01-27; Study Completion 2007-09-06

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital San Gerardo di Monza, University of Bicocca Monza, Milan, Italy